CLINICAL TRIAL: NCT03641495
Title: Effects of Pain Education and Therapeutic Exercise for Patients With Fibromyalgia
Brief Title: Pain Education and Therapeutic Exercise for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: University of Valladolid (Other)
Responsible Party: Principal Investigator, Sandra Jiménez, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Valladolid
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; therapeutic exercise; physiotherapy
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain education plus exercise therapy (PE + ET) (Experimental): Pain education according to the book "Explain Pain" written by Lorimer Moseley and David Butler
  Exercise therapy based primarily in aerobic exercise according clinical guidelines last recommendations.
  Interventions: Other: PE+ET
- Exercise therapy (ET) (Active Comparator): Exercise therapy based primarily in aerobic exercise according clinical guidelines last recommendations.
  Interventions: Other: ET

INTERVENTIONS:
Other: PE+ET — To explain the physiology of nervous system and the mechanism and modulation of acute and chronic pain.
  To perform different whole body aerobic exercises with a mild to moderate intensity according to Borg scale and maximum heart rate.
  Arms: Pain education plus exercise therapy (PE + ET)
Other: ET — To perform different whole body aerobic exercises with a mild to moderate intensity according to Borg scale and maximum heart rate.
  Arms: Exercise therapy (ET)

SUMMARY:
Fibromyalgia syndrome is characterized by chronic generalized musculoskeletal pain associated with fatigue, sleep disturbances and psychological problems. The European League Againts Rheumatism (EULAR) described an algorithm how to treat step by step these patients.

The objective of this trial is to evaluate if patient education plus therapeutic exercise is more effective in pain intensity, fatigue, function, strength, pain threshold, anxiety, depression, quality of life, quality of sleep, kinesiophobia, pain coping and biochemical and genetic markers and compared to therapeutic exercise.

For this purpose the investigators conduct a randomized controlled trial double-blind (patient and examiner). The investigators included patients diagnosed of fibromyalgia according to the American College of Rheumatology (ACR).

Patients included are randomized into 2 groups one receive education of pain neurophysiology plus exercise therapy and the other only exercise therapy. Groups receive 3 treatment sessions a week over 10 weeks.

The variables are measured at the beginning and end of treatment. And also some variables are measured before and after each session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed medically with Fibromyalgia
* Diagnosed according to the American College of Rheumatology criteria
* Agreement to attend to treatment sessions

Exclusion Criteria:

* Any kind of contraindications for physical activity
* Other kind of diseases that could limit the intervention
* Previous surgery last year
* Medication modifications in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity: VAS | Baseline
  The investigators measure the intensity of pain with a Visual Analogic Scale (VAS) pre-intervention at baseline
Pain Intensity: VAS | through study completion, an average 10 weeks
  The investigators measure the intensity of pain with a Visual Analogic Scale (VAS) at the end of the intervention
Fibromyalgia Impact Questionnaire | Baseline
  The investigators measure the impact of Fibromyalgia syndrome by Fibromyalgia Impact Questionnaire R (FIQ-R) pre-intervention at baseline
Fibromyalgia Impact Questionnaire | through study completion, an average 10 weeks
  The investigators measure the impact of Fibromyalgia syndrome by Fibromyalgia Impact Questionnaire R (FIQ-R) at the end of the intervention

SECONDARY OUTCOMES:
Fatigue | Baseline
  The investigators measure the fatigue with Multidimensional Fatigue Inventory (MFI-S) pre-intervention at baseline
Fatigue | through study completion, an average 10 weeks
  The investigators measure the fatigue with Multidimensional Fatigue Inventory (MFI-S) at the end of the intervention
Quality of Sleep | Baseline
  The investigators measure the quality of sleep with Pittsburg Sleeping Questionnaire Index (PSQI) at baseline
Quality of Sleep: Pittsburg Sleeping Questionnaire | through study completion, an average 10 weeks
  The investigators measure the quality of sleep with Pittsburg Sleeping Questionnaire Index (PSQI) at the end of the intervention
Functional Capacity | Baseline
  The investigators measure the functional capacity with Senior Fitness Test at baseline
Functional Capacity | through study completion, an average 10 weeks
  The investigators measure the functional capacity with Senior Fitness Test at the end of treatment
body strength | baseline
  The investigators measure the strength of arms with handgrip test, elbow flexion and knee extension with handheld dynamometer at baseline
body strength | through study completion, an average 10 weeks
  The investigators measure the strength of arms with handgrip test, elbow flexion and knee extension with handheld dynamometer at the end of treatment
Pressure pain threshold | baseline
  The investigators measure the pressure pain threshold of the 18 points described initially by the American College of rheumatology with a digital algometer at baseline
Pressure pain threshold | through study completion, an average 10 weeks
  The investigators measure the pressure pain threshold of the 18 points described initially by the American College of rheumatology with a digital algometer at the end of treatment
Anxiety and Depression | Baseline
  The investigators measure the anxiety and depression with Hospital Anxiety and Depression Scale (HADS) at baseline
Anxiety and Depression | through study completion, an average 10 weeks
  The investigators measure the anxiety and depression with Hospital Anxiety and Depression Scale (HADS) at the end of the intervention
kinesiophobia | baseline
  The investigators measure the kinesiophobia with TAMPA questionnaire at baseline
kinesiophobia | through study completion, an average 10 weeks
  The investigators measure the kinesiophobia with TAMPA questionnaire at the end of treatment
Quality of life: HAQ | baseline
  The investigators measure the quality of life with Health Assessment Questionnaire (HAQ) at baseline
Quality of life: HAQ | through study completion, an average 10 weeks
  The investigators measure the quality of life with ( Health Assessment Questionnaire (HAQ) at the end of treatment
Central sensitization | baseline
  The investigators measure the central sensitization with Chronic Pain Self-Efficacy Scale (CPSS) at baseline
Central sensitization | through study completion, an average 10 weeks
  The investigators measure the central sensitization with Chronic Pain Self-Efficacy Scale (CPSS) at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Jiménez del Barrio, Soria, Spain

IPD SHARING:
Plan to Share IPD: No
The patient data were confidential and were assigned a number to each patient to maintain confidentiality